CLINICAL TRIAL: NCT03091192
Title: A Phase III, Open Label, Randomised, Controlled, Multi-Centre Study To Assess the Efficacy and Safety of Savolitinib Versus Sunitinib in Patients With MET-Driven, Unresectable and Locally Advanced, Or Metastatic Papillary Renal Cell Carcinoma (PRCC)
Brief Title: Savolitinib vs. Sunitinib in MET-driven PRCC.
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: Hutchison Medipharma Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: D5082C00003; 2016-004108-73 (EudraCT Number)
Record Dates: First submitted 2017-02-09; First posted 2017-03-27 (Actual); Results first posted 2020-07-10 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Carcinoma; Carcinoma, Renal Cell; Kidney Neoplasms; Urologic Neoplasms; Kidney Diseases; Neoplasms by Site; Enzyme Inhibitors; Protein Kinase Inhibitors
Keywords: Papillary Renal Cell Cancer; AZD6094; Savolitinib
MeSH Terms: conditions — Carcinoma; Carcinoma, Renal Cell; Kidney Neoplasms; Urologic Neoplasms; Kidney Diseases; Neoplasms by Site | interventions — 1-(1-(imidazo(1,2-a)pyridin-6-yl)ethyl)-6-(1-methyl-1H-pyrazol-4-yl)-1H-(1,2,3)triazolo(4,5-b)pyrazine; Sunitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Savolitinib (Experimental): See: intervention description
  Interventions: Drug: Savolitinib
- Sunitinib (Active Comparator): See: intervention description
  Interventions: Drug: Sunitinib

INTERVENTIONS:
Drug: Savolitinib — 600 mg (400 mg if <50 kg) by mouth (PO) with a meal once daily (QD), continuously
  Other Names: AZD6094 (HMPL-504)/Volitinib
  Arms: Savolitinib
Drug: Sunitinib — 50 mg by mouth (PO) once daily (QD), with or w/o food, 4 weeks on/2weeks off
  Arms: Sunitinib

SUMMARY:
This study is designed for patients diagnosed with MET-driven, unresectable and locally advanced or metastatic Papillary Renal Cell Carcinoma. The purpose of this study is to see if an investigational new anti-cancer medication, savolitinib, is effective in treating patients with MET-driven PRCC, how it compares with another medication frequently used to treat this disease called sunitinib, and what side effects it might cause.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed PRCC, which is unresectable/locally advanced or metastatic with measurable disease as per RECIST 1.1. Patients with papillary urothelial carcinoma or renal pelvis cancer of the kidney are not considered PRCC and are not eligible.
2. Confirmation of MET-driven PRCC without co-occurring FH or VHL mutations from an FFPE tumour sample using the sponsor-designated central laboratory validated NGS assay
3. Patients who have received no prior systemic therapy as well as those who have received prior systemic therapy for PRCC in the advanced setting.* Patients can be treatment-naïve, or previously treated, but cannot have previously received sunitinib or a MET inhibitor. Patients who have received prior systemic therapy must have had disease progression in soft tissue disease or bone within 6 months of the last dose of the most recent systemic therapy
4. Adequate haematological, renal, cardiac and liver functions
5. Karnofsky performance status ≥ 80

Exclusion Criteria:

1. Most recent cytotoxic chemotherapy, immunotherapy, chemo-immunotherapy, or investigational agents <28 days from the date of randomisation. Most recent non cytotoxic targeted therapy <14 days from the date of randomisation.
2. Prior treatment with a MET inhibitor (e.g. foretinib, crizotinib, cabozantinib, onartuzumab or previous savolitinib) or sunitinb.
3. Treatment with strong inducers or inhibitors of CYP3A4 or strong inhibitors of CYP1A2, taken within 2 weeks or not possible to be stopped for at least 2 week before the date of randomisation. Herbal medications cannot be taken within 7 days of the date of randomisation (3 weeks for St John's wort).
4. Wide field radiotherapy administered ≤28 days or limited field radiation for palliation ≤7 days prior to the date of randomisation
5. Major surgical procedures ≤28 days of randomisation or minor surgical procedures ≤7 days. No waiting is required following port-a-cath placement.
6. Previously untreated brain metastases
7. Serious active infection or gastrointestinal disease
8. Presence of other active cancers, or history of treatment for invasive cancer within the last 5 years.
9. Mean resting QTcF >470 msec for women and >450 msec for men on the Part 2 screening triplicate ECGs or factors that may increase the risk of QTcF prolongation such as chronic hypokalaemia not correctable with supplements, congenital or familial long QT syndrome, or family history of unexplained sudden death under 40 years of age in first-degree relatives or any concomitant medication known to prolong the QT interval and cause Torsades de Pointes

Ages: 18 Years to 130 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2017-07-25 (Actual); Primary Completion 2019-08-18 (Actual); Study Completion 2026-12-31 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Toni K Choueiri, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (45):
- United States (8):
  - Research Site, La Jolla, California
  - Research Site, Atlanta, Georgia
  - Research Site, Chicago, Illinois
  - Research Site, Iowa City, Iowa
  - Research Site, Boston, Massachusetts
  - Research Site, Kansas City, Missouri
  - Research Site, New York, New York
  - Research Site, Nashville, Tennessee
- Brazil (8):
  - Research Site, Barretos
  - Research Site, Curitiba
  - Research Site, Passo Fundo
  - Research Site, Pelotas
  - Research Site, Porto Alegre
  - Research Site, Rio de Janeiro
  - Research Site, São José do Rio Preto
  - Research Site, São Paulo
- France (3):
  - Research Site, Bordeaux
  - Research Site, Vandœuvre-lès-Nancy
  - Research Site, Villejuif
- Italy (7):
  - Research Site, Arezzo
  - Research Site, Meldola
  - Research Site, Milan
  - Research Site, Modena
  - Research Site, Orbassano
  - Research Site, Pavia
  - Research Site, Roma
- Russia (8):
  - Research Site, Krasnoyarsk
  - Research Site, Moscow
  - Research Site, Murmansk
  - Research Site, Nizhny Novgorod
  - Research Site, Obninsk
  - Research Site, Omsk
  - Research Site, Saint Petersburg
  - Research Site, Volgograd
- South Korea (5):
  - Research Site, Daejeon
  - Research Site, Goyang-si
  - Research Site, Hwasun-gun
  - Research Site, Incheon
  - Research Site, Seoul
- Ukraine (6):
  - Research Site, Dnipro
  - Research Site, Ivano-Frankivsk
  - Research Site, Kharkiv Region
  - Research Site, Kyiv
  - Research Site, Odesa
  - Research Site, Sumy

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All request will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
  Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the de-identified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- [Derived] Choueiri TK, Heng DYC, Lee JL, Cancel M, Verheijen RB, Mellemgaard A, Ottesen LH, Frigault MM, L'Hernault A, Szijgyarto Z, Signoretti S, Albiges L. Efficacy of Savolitinib vs Sunitinib in Patients With MET-Driven Papillary Renal Cell Carcinoma: The SAVOIR Phase 3 Randomized Clinical Trial. JAMA Oncol. 2020 Aug 1;6(8):1247-1255. doi: 10.1001/jamaoncol.2020.2218. PMID 32469384
- [Derived] Maia MC, Salgia M, Pal SK. Harnessing cell-free DNA: plasma circulating tumour DNA for liquid biopsy in genitourinary cancers. Nat Rev Urol. 2020 May;17(5):271-291. doi: 10.1038/s41585-020-0297-9. Epub 2020 Mar 17. PMID 32203306
- See also: Related Info — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D5082C00003&attachmentIdentifier=0584547a-9e19-4f7a-b5dc-e8c54e51e817&fileName=d5082c00003-csp-v6-redacted_-_CTT_pdfa.pdf&versionIdentifier=
- See also: Related Info — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D5082C00003&attachmentIdentifier=e4538a3c-36dc-470a-9f66-b4109d935ae7&fileName=d5082c00003-sap-ed-2-redacted-CTT_pdfa.pdf&versionIdentifier=

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First subject enrolled: 25 July 2017. Last subject last visit: 18 August 2019. Data cut off: 19 August 2019. The study was terminated prematurely. Randomized subjects continue to receive IMP as clinically indicated by PI; safety information is being collected for those subjects.
Groups:
- Savolitinib QD: Savolitinib QD
- Sunitinib QD: Sunitinib QD
Period: Overall Study
Arm/Group | Savolitinib QD | Sunitinib QD
Started | 33 | 27
Completed | 0 | 0
Not Completed | 33 | 27
Not completed — Study terminated by sponsor | 21 | 14
Not completed — Death | 9 | 13
Not completed — Withdrawal by Subject | 2 | 0
Not completed — Lost to Follow-up | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Savolitinib QD | Sunitinib QD | Total
Number analyzed (Participants) | 33 | 27 | 60
Age, Continuous [Mean (Standard Deviation); unit: Years] | 56.7 (13.81) | 63.1 (9.60) | 59.6 (12.43)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 10 | 14
  Male | 29 | 17 | 46
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 3 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 1 | 2
  White | 29 | 23 | 52
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival (PFS) by Blinded Independent Central Review (BICR)
Description: Per Response Evaluation Criteria in Solid Tumours (RECIST v1.1) assessed by MRI or CT: Progressive Disease (PD): >= 20% increase in the sum of diameters of TLs and an absolute increase in sum of diameters of >=5mm (compared to the previous minimum sum) or progression of NTLs or a new lesion. PFS is the time from date of randomisation until the date of PD (defined by Recist 1.1 and confirmed by BICR) or death (by any cause in the absence of progression) regardless of whether the patient withdrew from randomised therapy or received another anti-cancer therapy prior to progression.
Time Frame: RECIST tumour assessments every 6 weeks from randomisation until disease progression as defined by Recist 1.1 and confirmed by BICR.
Population: Full Analysis Set (All randomised patients)
Measure: Median (95% Confidence Interval); unit: Months
Units Other Than Participants: Events
Arm/Group | Savolitinib QD | Sunitinib QD
Number analyzed (Participants) | 33 | 27
Number analyzed (Events) | 17 | 20
Months | 7.0 [2.8 to NA] — The upper limit was not calculable. | 5.6 [4.1 to 6.9]
Statistical Analysis 1: Comparison: Savolitinib QD vs Sunitinib QD; Test type: Superiority; p = 0.313, Log Rank; Hazard Ratio (HR) = 0.71, 95% CI 2-sided [0.37 to 1.36]

2. Secondary Outcome: Overall Survival (OS)
Description: Time between the date of randomisation and the date of death due to any cause.
Time Frame: as for outcome 1
Population: Full Analysis Set (All randomised patients)
Measure: Count of Participants; unit: Participants
Arm/Group | Savolitinib QD | Sunitinib QD
Number analyzed (Participants) | 33 | 27
Participants
  Died | 9 | 13
  Terminated study prior to death | 24 | 14
Statistical Analysis 1: Comparison: Savolitinib QD vs Sunitinib QD; Test type: Superiority; p = 0.110, Log Rank; Hazard Ratio (HR) = 0.51, 95% CI 2-sided [0.21 to 1.17] — A hazard ratio < 1 favours Savolitinib

3. Secondary Outcome: Objective Response Rate (ORR) by BICR
Description: Per Response Evaluation Criteria in Solid Tumours (RECIST v1.1) assessed by MRI or CT: Complete Response (CR): Disappearance of all target and non-target lesions and no new lesions; Partial Response (PR): >= 30% decrease in the sum of diameters of Target Lesions (compared to baseline) and no new lesions. ORR is the percentage of patients with at least 1 visit response of CR or PR prior to progression or any further therapy.
Time Frame: as for outcome 1
Population: Full Analysis Set (All randomised patients)
Measure: Number (95% Confidence Interval); unit: % of participants
Arm/Group | Savolitinib QD | Sunitinib QD
Number analyzed (Participants) | 33 | 27
% of participants | 27.3 [13.3 to 45.5] | 7.4 [0.9 to 24.3]

4. Secondary Outcome: Duration of Response (DoR) by BICR
Description: Per Response Evaluation Criteria in Solid Tumours (RECIST v1.1) assessed by MRI or CT: Complete Response (CR): Disappearance of all target and non-target lesions and no new lesions; Partial Response (PR): >= 30% decrease in the sum of diameters of Target Lesions (compared to baseline) and no new lesions. DoR is the time from the date of first documented response until the date of documented progression or death in the absence of disease progression.
Time Frame: as for outcome 1
Population: Duration of Response (DoR) by BICR was calculated for all responders (N=11)
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Savolitinib QD | Sunitinib QD
Number analyzed (Participants) | 9 | 2
Months | NA [NA to NA] — There were no patients (0/9) with an objective response who subsequently had PFS events. There were 2 subjects that are known to have died but are censored for PFS as death occurred > 14 weeks after last evaluable RECIST assessment. | 8.3 [NA to NA] — The confidence limits were not calculable. There was 1 patient with an objective response who subsequently progressed or died in the sunitinib group.

5. Secondary Outcome: Disease Control Rate (DCR) at 6 Months by BICR
Description: Disease control rate at 6 months is defined as the percentage of patients who have a best objective response of Complete Response or Partial Response in that period or who have demonstrated Stable Disease for a minimum interval of 23 weeks.
Time Frame: as for outcome 1
Population: Full Analysis Set (All randomised patients)
Measure: Number (95% Confidence Interval); unit: % of participants
Arm/Group | Savolitinib QD | Sunitinib QD
Number analyzed (Participants) | 33 | 27
% of participants | 48.5 [30.8 to 66.5] | 37.0 [19.4 to 57.6]

6. Secondary Outcome: Disease Control Rate (DCR) at 12 Months by BICR
Description: Disease control rate at 12 months is defined as the percentage of patients who have a best objective response of complete responses or partial responses in that period or who have demonstrated stable disease for a minimum interval of 47 weeks.
Time Frame: as for outcome 1
Population: Full Analysis Set (All randomised patients)
Measure: Number (95% Confidence Interval); unit: % of participants
Arm/Group | Savolitinib QD | Sunitinib QD
Number analyzed (Participants) | 33 | 27
% of participants | 30.3 [15.6 to 48.7] | 22.2 [8.6 to 42.3]

ADVERSE EVENTS:
Time Frame: Adverse Events (AEs) and Serious Adverse Events (SAEs) were collected throughout the study, from date of informed consent until 30 days after the last dose of study treatment.
Description: Systematic assessment due to regular investigator assessment at study visits.
Arm/Group | Savolitinib QD | Sunitinib QD
All-Cause Mortality (participants affected / at risk) | 9/33 | 13/27
Serious Adverse Events (participants affected / at risk) | 8/33 | 8/27
Other Adverse Events (participants affected / at risk) | 25/33 | 27/27
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Savolitinib QD (N=33) | Sunitinib QD (N=27)
Pneumonia (Infections and infestations) | 1 (1) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Drug hypersensitivity (Immune system disorders) | 1 (1) | 0 (0)
Thrombotic cerebral infarction (Nervous system disorders) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac failure (Cardiac disorders) | 0 (0) | 1 (1)
Myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1)
Ventricular tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Hypertensive urgency (Vascular disorders) | 0 (0) | 1 (1)
Thrombophlebitis (Vascular disorders) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Anal fistula (Gastrointestinal disorders) | 0 (0) | 1 (1)
Ascites (Gastrointestinal disorders) | 1 (1) | 0 (0)
Incarcerated umbilical hernia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Biliary dilatation (Hepatobiliary disorders) | 1 (1) | 0 (0)
Cholangitis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Jaundice (Hepatobiliary disorders) | 1 (1) | 0 (0)
Condition aggravated (General disorders) | 0 (0) | 1 (1)
Oedema peripheral (General disorders) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 1 (1) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Savolitinib QD (N=33) | Sunitinib QD (N=27)
Conjuntivitis (Infections and infestations) | 0 (0) | 2 (2)
Urinary tract infection (Infections and infestations) | 0 (0) | 4 (4)
Anaemia (Blood and lymphatic system disorders) | 2 (2) | 12 (18)
Leukopenia (Blood and lymphatic system disorders) | 1 (1) | 2 (3)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 5 (11)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 6 (8)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 8 (10)
Dyslipidaemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Hyperglycaemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 3 (3) | 2 (2)
Dysgeusia (Nervous system disorders) | 0 (0) | 2 (2)
Headache (Nervous system disorders) | 3 (3) | 4 (4)
Taste disorder (Nervous system disorders) | 0 (0) | 2 (3)
Tachycardia (Cardiac disorders) | 2 (2) | 1 (1)
Capillary leak syndrome (Vascular disorders) | 3 (3) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 6 (9)
Cough (Respiratory, thoracic and mediastinal disorders) | 4 (5) | 6 (6)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 7 (7) | 4 (4)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 4 (4)
Constipation (Gastrointestinal disorders) | 2 (2) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 6 (19)
Dyspepsia (Gastrointestinal disorders) | 1 (2) | 3 (3)
Nausea (Gastrointestinal disorders) | 2 (3) | 9 (13)
Odynophagia (Gastrointestinal disorders) | 0 (0) | 2 (2)
Stomatitis (Gastrointestinal disorders) | 1 (1) | 2 (2)
Vomiting (Gastrointestinal disorders) | 1 (1) | 4 (6)
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 (0) | 7 (7)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2)
Rash (Skin and subcutaneous tissue disorders) | 2 (3) | 1 (1)
Yellow skin (Skin and subcutaneous tissue disorders) | 0 (0) | 4 (4)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (3) | 2 (4)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 5 (5)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (2) | 3 (4)
Chronic kidney disease (Renal and urinary disorders) | 2 (2) | 1 (1)
Proteinuria (Renal and urinary disorders) | 1 (1) | 2 (2)
Asthenia (General disorders) | 1 (1) | 5 (5)
Face oedema (General disorders) | 0 (0) | 3 (3)
Fatigue (General disorders) | 2 (2) | 5 (5)
Mucosal inflammation (General disorders) | 0 (0) | 3 (4)
Oedema peripheral (General disorders) | 11 (17) | 3 (4)
Peripheral swelling (General disorders) | 2 (2) | 0 (0)
Pyrexia (General disorders) | 2 (2) | 2 (2)
Alanine aminotransferase increased (Investigations) | 7 (11) | 3 (5)
Amylase increased (Investigations) | 1 (1) | 2 (2)
Aspartate aminotransferase increased (Investigations) | 7 (9) | 5 (7)
Blood creatinine increased (Investigations) | 9 (10) | 2 (2)
Blood thyroid stimulating hormone decreased (Investigations) | 0 (0) | 3 (3)
Blood thyroid stimulating hormone increased (Investigations) | 0 (0) | 4 (7)
Body temperature increased (Investigations) | 3 (3) | 2 (2)
Ejection fraction decreased (Investigations) | 0 (0) | 3 (3)
Lipase increased (Investigations) | 0 (0) | 2 (2)
Neutrophil count decreased (Investigations) | 0 (0) | 5 (11)
Platelet count decreased (Investigations) | 1 (2) | 4 (5)
Thyroxine increased (Investigations) | 0 (0) | 2 (2)
Weight decreased (Investigations) | 0 (0) | 2 (2)
White blood cell count decreased (Investigations) | 1 (1) | 3 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2018-12-19): https://cdn.clinicaltrials.gov/large-docs/92/NCT03091192/Prot_004.pdf
  • Statistical Analysis Plan (2019-08-28): https://cdn.clinicaltrials.gov/large-docs/92/NCT03091192/SAP_000.pdf